CLINICAL TRIAL: NCT01815138
Title: A Prospective Double-blind Randomized Trial Comparing Pregnancy Rates After Low Dose Human Chorionic Gonadotropin (hCG) at the Time of Gonadotropin Releasing Hormone (GnRH) Agonist Trigger or 35 Hours Later for the Prevention of OHSS
Brief Title: Co-administration of Low Dose hCG at the Time of GnRH Agonist Trigger or 35 Hours Later for the Prevention of OHSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lawrence Engmann, MD, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-098-3
Record Dates: First submitted 2013-03-16; First posted 2013-03-20 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS, GnRH agonist trigger, low dose hCG, PCOS, IVF
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome; Polycystic Ovary Syndrome | interventions — Chorionic Gonadotropin; Profasi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hCG given at time of GnRHa trigger (Experimental): Adjuvant low dose hCG 1,000 IU administered at the time of GnRH agonist trigger.
  Placebo administered 35 hours after GnRH agonist trigger
  Interventions: Drug: hCG
- hCG given 35 hours after GnRHa trigger (Active Comparator): Placebo administered at the time of GnRH agonist trigger
  Adjuvant low dose hCG 1,500 IU administered 35 hours after GnRH agonist trigger.
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG — Adjuvant low dose hCG 1,000 IU administered at the time of GnRH agonist trigger
  Other Names: Pregnyl, Profasi
  Arms: hCG given at time of GnRHa trigger
Drug: hCG — Adjuvant low dose hCG 1,500 IU administered 35 hours after GnRH agonist trigger
  Other Names: Pregnyl, Profasi
  Arms: hCG given 35 hours after GnRHa trigger

SUMMARY:
This a prospective randomized double blind study involving patients at high risk of OHSS development with peak serum E2 levels < 4,000 pg/ml comparing the ongoing pregnancy rates in patients who receive adjuvant hCG 1,000 IU at the time of GnRH agonist trigger or adjuvant hCG 1,500 IU 35 hours after GnRH agonist trigger.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is an iatrogenic complication of controlled ovarian hyperstimulation which may result in significant morbidity and rarely mortality as well as significant financial and psychological distress. GnRH agonist trigger has been shown to be effective in OHSS prevention. However, the adoption of its use has not been widely accepted in view of concerns regarding potential impairment of implantation.

Intensive luteal phase supplementation with estrogen (E2) and progesterone (P) is important due to the strong evidence of abnormal luteal phase serum E2 and P profiles. However, it has been shown that optimal conception rates is not achieved for high risk patients with peak serum E2 < 4,000 pg/ml despite aggressive steroidal supplementation. It has been proposed that the use of adjuvant low dose hCG at the time of GnRH agonist trigger or 35 hours later will rescue some of the corpora lutea and help improve corpora lutea function and improve pregnancy rates.

The study will evaluate patients at high risk of OHSS development with peak serum E2 < 4,000 pg/mL to determine whether timing of low dose hCG administration affects ongoing pregnancy rates or risk of OHSS. Markers of corpus luteum function such as serum 17 hydroxy-progesterone and prorenin during the luteal phase and early pregnancy will help elucidate further the effect of adjuvant low dose hCG with GnRH agonist trigger on corpus luteum function.

ELIGIBILITY:
Inclusion Criteria:

* Normal baseline serum follicle stimulating hormone, polycystic ovarian syndrome (PCOS), Polycystic ovarian morphology, Previous high responder or previous OHSS, must have > 14 follicles of over 11 mm in diameter and with peak serum E2 levels < 4,000 pg/mL on the day of trigger of oocyte maturation.

Exclusion Criteria:

* Hypothalamic dysfunction, Patients with < 14 follicles < 11 mm in diameter, peak serum E2 levels >= 4,000 pg/mL.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Engmann, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Griffin D, Benadiva C, Kummer N, Budinetz T, Nulsen J, Engmann L. Dual trigger of oocyte maturation with gonadotropin-releasing hormone agonist and low-dose human chorionic gonadotropin to optimize live birth rates in high responders. Fertil Steril. 2012 Jun;97(6):1316-20. doi: 10.1016/j.fertnstert.2012.03.015. Epub 2012 Apr 3. PMID 22480822
- [Background] Kummer N, Benadiva C, Feinn R, Mann J, Nulsen J, Engmann L. Factors that predict the probability of a successful clinical outcome after induction of oocyte maturation with a gonadotropin-releasing hormone agonist. Fertil Steril. 2011 Jul;96(1):63-8. doi: 10.1016/j.fertnstert.2011.04.050. Epub 2011 May 12. PMID 21565337
- [Background] Engmann L, DiLuigi A, Schmidt D, Nulsen J, Maier D, Benadiva C. The use of gonadotropin-releasing hormone (GnRH) agonist to induce oocyte maturation after cotreatment with GnRH antagonist in high-risk patients undergoing in vitro fertilization prevents the risk of ovarian hyperstimulation syndrome: a prospective randomized controlled study. Fertil Steril. 2008 Jan;89(1):84-91. doi: 10.1016/j.fertnstert.2007.02.002. Epub 2007 Apr 26. PMID 17462639
- [Background] Humaidan P. Luteal phase rescue in high-risk OHSS patients by GnRHa triggering in combination with low-dose HCG: a pilot study. Reprod Biomed Online. 2009 May;18(5):630-4. doi: 10.1016/s1472-6483(10)60006-5. PMID 19549440
- [Background] Humaidan P, Bungum L, Bungum M, Yding Andersen C. Rescue of corpus luteum function with peri-ovulatory HCG supplementation in IVF/ICSI GnRH antagonist cycles in which ovulation was triggered with a GnRH agonist: a pilot study. Reprod Biomed Online. 2006 Aug;13(2):173-8. doi: 10.1016/s1472-6483(10)60612-8. PMID 16895629
- [Derived] Kaye L, Griffin D, Thorne J, Neuber E, Nulsen J, Benadiva C, Engmann L. Independent serum markers of corpora lutea function after gonadotropin-releasing hormone agonist trigger and adjuvant low dose human chorionic gonadotropin in in vitro fertilization. Fertil Steril. 2019 Sep;112(3):534-544. doi: 10.1016/j.fertnstert.2019.04.034. Epub 2019 Jun 18. PMID 31227286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients that met initial study criteria were enrolled and consented before starting ovarian stimulation. Final randomization occurred during stimulation. Therefore patients who were enrolled and consented may drop out before randomization, either because they did not meet the final inclusion criteria in did not undergo IVF.
Groups:
- hCG Given at Time of GnRHa Trigger: Adjuvant low dose hCG 1,000 IU administered at the time of GnRH agonist trigger.
  Placebo administered 35 hours after GnRH agonist trigger
  hCG: Adjuvant low dose hCG 1,000 IU administered at the time of GnRH agonist trigger
- hCG Given 35 Hours After GnRHa Trigger: Placebo administered at the time of GnRH agonist trigger
  Adjuvant low dose hCG 1,500 IU administered 35 hours after GnRH agonist trigger.
  hCG: Adjuvant low dose hCG 1,500 IU administered 35 hours after GnRH agonist trigger
Period: Overall Study
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
Started | 34 | 37
Completed | 26 | 31
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger | Total
Number analyzed (Participants) | 26 | 31 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (3.3) | 32.2 (3.4) | 31.8 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 57
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: "kg/m^2"] | 26.3 (4.8) | 27.4 (5.5) | 26.9 (5.2)
Anti Mullerian Hormone (AMH) [Mean (Standard Deviation); unit: ng/ml] | 8.3 (5.8) | 8.4 (4.9) | 8.35 (5.2)
Follicle Stimulating Hormone (FSH) [Mean (Standard Deviation); unit: IU/L] | 5.6 (1.7) | 5.2 (1.6) | 5.5 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy
Description: Positive serum pregnancy test and ultrasound evidence of fetal pole and fetal heart rate .
Time Frame: Through time of study completion, on average 1-2years
Population: per protocol analysis
Measure: Number; unit: participants
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
Number analyzed (Participants) | 26 | 31
participants | 15 | 19

2. Secondary Outcome: Ovarian Hyperstimulation Syndrome
Description: Evaluation of symptoms and signs of OHSS at 9 days after trigger of oocyte maturation. Patients who also present with symptoms of OHSS wil also be evaluated for OHSS within 4 weeks after oocyte maturation.
Time Frame: Within 4 weeks of oocyte retrieval
Population: Women with normal or high response to IVF, peak estradiol on day of trigger less than 4000 pg/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
Number analyzed (Participants) | 26 | 31
Participants | 1 | 3
Statistical Analysis 1: Comparison: hCG Given at Time of GnRHa Trigger vs hCG Given 35 Hours After GnRHa Trigger; Test type: Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.05

3. Other Pre Specified Outcome: Markers of Corpus Luteum Function
Description: A subset of patients (20 patients in each group) will have serum frozen for subsequent analysis of 17 hydroxy progesterone and prorenin.
Time Frame: Within 60 days after trigger of oocyte maturation
Population: Subset of women included in larger study, normal or high responders, peak estradiol level less than 4000 pg/mL on day of trigger.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
Number analyzed (Participants) | 10 | 20
ng/mL
  Early luteal 17-OH-Progesterone | 13.68 (11.0) | 21.77 (8.5)
  Day 16 Prorenin | 1.13 (0.8) | 2.22 (1.6)
Statistical Analysis 1: Comparison: hCG Given at Time of GnRHa Trigger vs hCG Given 35 Hours After GnRHa Trigger; Test type: Superiority; p = 0.04, t-test, 2 sided

4. Other Pre Specified Outcome: Proportion of Patients With Abdominal Distension
Description: Patients will complete a questionnaire to determine if there is a difference in the effect of the intervention on the quality of life (abdominal distension) of the patients from the day of trigger of oocyte maturation until menses or positive pregnancy test.
Time Frame: Within 2 weeks after trigger of oocyte maturation
Population: Some patients did not complete the questionnaire. Abdominal distension analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
Number analyzed (Participants) | 20 | 27
Participants
  Abdominal distension | 2 | 11
  abdominal pain | 1 | 9

ADVERSE EVENTS:
Arm/Group | hCG Given at Time of GnRHa Trigger | hCG Given 35 Hours After GnRHa Trigger
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/31
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCG Given at Time of GnRHa Trigger (N=26) | hCG Given 35 Hours After GnRHa Trigger (N=31)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Patient diagnosed with un-ruptured ectopic pregnancy and required a laparoscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No